CLINICAL TRIAL: NCT05117827
Title: Pediatric Powered Wheelchair Standing Devices: An Exploratory Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grand Valley State University (Other)
Responsible Party: Principal Investigator, Lisa Kenyon, Professor, Grand Valley State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-052-H
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy; Spinal Muscular Atrophy; Spinal Cord Injuries; Spina Bifida; Development Delay; Genetic Disease
MeSH Terms: conditions — Cerebral Palsy; Muscular Atrophy, Spinal; Spinal Cord Injuries; Spinal Dysraphism; Learning Disabilities; Genetic Diseases, Inborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Power Wheelchair Standing Device User (Experimental)
  Interventions: Device: Power Wheelchair Standing Device

INTERVENTIONS:
Device: Power Wheelchair Standing Device — A power wheelchair standing device is a power wheelchair that allows a child to electronically move between sitting and standing. It can be driven in either position. The Permobil F5 Corpus VS is the specific power wheelchair standing device to be used in this study.

SUMMARY:
For children who use a power wheelchair, a powered wheelchair standing device (PWSD) may be considered for daily use. A PWSD allows a child to electronically move between sitting and standing and can be driven in either position. Existing published PWSD research in pediatrics is limited to boys with Duchenne muscular dystrophy (DMD).(1, 2) While these studies provide some insights into PWSD use in boys with DMD, they do not reflect PWSD use in children with other conditions. The purpose of this exploratory study is to determine the feasibility of a research protocol exploring use of a PWSD in children who have neurodevelopmental conditions other than DMD.

ELIGIBILITY:
Inclusion Criteria:

1. Is 5-17 years of age. NOTE: Participants must be under 18 for the duration of the study.
2. Diagnosed with a neurodevelopmental condition resulting in an inability to functionally ambulate.
3. Can safely assume and maintain a supported standing position
4. Has sufficient upper extremity and function to safely use a PWSD
5. Can communicate pain or discomfort through verbalization, vocalization, use of augmented communication, etc.
6. Can safely use the PWSD in areas of their home
7. Has at least one parent/caregiver who is able to converse in English and actively participate in a device-use education provided in English
8. The PerMobil PWSD can be set up to meet the child's specific needs
9. Medical Clearance to trial the PWSD
10. Participants must reside in Michigan

Exclusion Criteria:

1. Has a diagnosis of Duchenne muscular dystrophy.
2. Any reason that it would not be safe for the child to use a PWSD

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Participation in children | 2 years
  Does using a PWSD increase participation in children who have neurodevelopmental conditions other than DMD?

SECONDARY OUTCOMES:
Parental/caregiver perceptions | 2 years
  Does using a PWSD influence parental/caregiver perceptions of their child's emotional/behavioral status?
Children's perceptions | 2 years
  For children who are able to respond to questions and participate in an interview using either verbal or augmented communication, does using a PWSD influence their own perceptions of their emotional/behavioral status?

CONTACTS AND LOCATIONS:
Locations (1):
- Grand Valley State University, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team may share research data related to study outcomes from this study with other investigators. If this occurs, the data will not contain identifiable data.
Supporting Information: Study Protocol
Time Frame: 2 years
Access Criteria: Contact PI